CLINICAL TRIAL: NCT01929304
Title: Assessment of Patient Understanding and Preference of Rescue Venous Access When Shown a Narrated Video Vignette Versus Traditional Paper Information Sheet
Brief Title: Difficult Intravenous Access Perception: Difficult IV Access - Assessment of Patient Understanding
Acronym: DIVA
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 818394b
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Understanding Emergency Room Procedures
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Video: Patients in this group will be shown an informational video, narrated in English.
  Interventions: Other: Survey
- Text: Patients in this group will read a single-page printed information sheet in English.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey
  Other Names: Patients will complete a survey to assess their understanding and preferences.

SUMMARY:
Aim: Patient Perception: This aim broadly intends to use traditional script versus a brief video education vignette to determine understanding and preferences among general emergency department patients of rescue access techniques. A challenge of emergency care is providing patient education surrounding procedures in a standardized and patient-oriented manner. This data would provide insight on a patient's understanding of the risks and benefits of rescue access, assess patient preference, and potentially influence what rescue technique is employed in the future. This information may also give us insight onto why DIVA patients might refuse randomization.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 18 years of age
* fluent in English
* hemodynamically stable emergency department patient

Exclusion Criteria:

* history of or current status of difficult intravenous access

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible for enrollment would be any hemodynamically stable adult 18 years of age or older who is a HUP Emergency Department patient, able to provide informed consent, without history of difficult intravenous access, and able to speak, read, hear, and speak English fluently.
Sampling Method: Non-Probability Sample
Enrollment: 1180 (Actual)
Dates: Start 2013-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Patient Understanding | Baseline
  Assess patients' understanding of and preferences regarding emergency department procedures: ultrasound-guided IV access and intra-osseous access.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States